CLINICAL TRIAL: NCT02347293
Title: Indigestible Carbohydrates in an Over-night Design as Means to Modulate Colonic Events, With Specific Focus on Metabolism and Satiety
Brief Title: Over-night Effect of Dietary Fiber on Glucose Metabolism and Satiety
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Jonna Sandberg, MSc, postgraduate student, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr2013/241b
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- + ind. CHO (Experimental): Test meals: intake of high levels of indigestible carbohydrates the evening prior to measurements of variables
  Interventions: Other: High levels of indigestible carbohydrates
- - ind. CHO (Experimental): Reference meal: scarce intake of indigestible carbohydrates the evening prior to measurements of variables
  Interventions: Other: Low levels of indigestible carbohydrates

INTERVENTIONS:
Other: High levels of indigestible carbohydrates
  Arms: + ind. CHO
Other: Low levels of indigestible carbohydrates
  Arms: - ind. CHO

SUMMARY:
The experimental model is a semi-acute, over-night, study where the purpose is to evaluate food factors related to colonially derived regulation and satiety in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normal fasting blood glucose
* BMI 19-25 kg/m2

Exclusion Criteria:

* Gastrointestinal diseases
* Food allergies e.g. lactose-, gluten intolerance
* Metabolic disorder e.g. diabetes
* Tobacco/snuff users
* No antibiotic or probiotic intake 2 weeks prior and during study.
* Vegetarians

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Blood Glucose, levels of glucose in blood | Postprandial 0-180 min after breakfast
Insulin, levels of insulin in blood | Postprandial 0-180 min after breakfast
Appetite hormones, levels of Peptide YY (PYY) in blood | Postprandial 0-180 min after breakfast
Markers of colonic fermentation, levels of hydrogen in breath | Postprandial 0-180 min after breakfast
Inflammation markers, levels of Interleukin-6 (IL-6) in blood | Postprandial 0-180 min after breakfast

SECONDARY OUTCOMES:
Subjective satiety, as measured by VAS | Postprandial 0-180 min after breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, PhD, Principal Investigator — Lund University
Locations (1):
- Medicon Village, Lund, Sweden

REFERENCES:
- [Derived] Gyll J, Ridell K, Ohlund I, Karlsland Akeson P, Johansson I, Lif Holgerson P. Vitamin D status and dental caries in healthy Swedish children. Nutr J. 2018 Jan 16;17(1):11. doi: 10.1186/s12937-018-0318-1. PMID 29338758
- [Derived] Sandberg JC, Bjorck IME, Nilsson AC. Effects of whole grain rye, with and without resistant starch type 2 supplementation, on glucose tolerance, gut hormones, inflammation and appetite regulation in an 11-14.5 hour perspective; a randomized controlled study in healthy subjects. Nutr J. 2017 Apr 21;16(1):25. doi: 10.1186/s12937-017-0246-5. PMID 28431559